CLINICAL TRIAL: NCT02289040
Title: A Feasibility Study to Consider the Role of Microvesicles (MV) and MV Derived microRNA (miRNA) in Acute Kidney Injury (AKI) Following Paediatric Cardiac Surgery: p-MiVAKI Study
Brief Title: Acute Kidney Injury Following Paediatric Cardiac Surgery
Acronym: p-MiVAKI
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); Heart Link Children's Charity (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0463; 14/EM/1136 (Other: East Midlands - Nottingham 1 Research Ethics Committee)
Record Dates: First submitted 2014-09-02; First posted 2014-11-13 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2017-05

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Microvesicles; microRNA; Paediatric cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * serum
  * EDTA plasma
  * citrated blood
  * hirudin blood
  * urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children undergoing cardiac surgery: Paediatric patients (<17 years with a body weight >2000g) undergoing cardiac surgery for congenital heart disease with extracorporeal circulation
  Interventions: Procedure: cardiac surgery

INTERVENTIONS:
Procedure: cardiac surgery — cardiac surgery with extracorporeal circulation for congenital heart disease

SUMMARY:
Acute kidney injury (AKI) complicates over 50% of cardiac surgical procedures in children where it increases morbidity and the use of healthcare resources. The pathogenesis of AKI is poorly understood, current diagnostic tests lack specificity and sensitivity, and there is no effective treatment. Improving outcomes in patients at risk of AKI has recently been defined as a National Health Service priority. The investigators are currently undertaking a program of work that is evaluating the role of plasma-derived microvesicles (MV) and MV associated microRNAs (miRNA) as diagnostic biomarkers or therapeutic targets in cardiac surgery patients at risk of developing AKI. Preliminary results indicate that these biomarkers may have clinical utility in adults. An important consideration is whether these biomarkers also have utility in children undergoing cardiac surgery. Measurement of MV at serial time points in children presents ethical challenges related to conducting clinical research in critically ill subjects. It also presents technical challenges related to the very small volumes of blood that may be sampled safely from babies and infants undergoing surgery. The aim of the study is to provide estimates of the perioperative variance of MV concentrations in 24 children undergoing cardiac surgery, as well as the frequency of AKI and other adverse events, protocol adherence and recruitment rates. This will assist with the design of a subsequent prospective observational study that will consider the role of MV/miRNA in children undergoing cardiac surgery.

DETAILED DESCRIPTION:
This is a prospective, single-centre observational feasibility study that will measure changes in MV signalling and their relationship to inflammatory responses after cardiac surgery in children.

The investigators primary hypothesis is that inflammatory renal injury following paediatric cardiac surgery is regulated by circulating MV and more specifically MV associated miRNA.

The investigators secondary hypotheses are:

1. MV derived signals will differ in cyanotic patients, a patient group at significantly increased risk for AKI.
2. MV subsets and/or MV derived miRNA may act as novel diagnostic biomarkers for AKI.

To assist with the design of a prospective observational study that will test these hypotheses the investigators propose to undertake a feasibility study in 24 children. The objectives of this feasibility study are:

A.To establish the numbers of patients that are eligible for enrolment in the study, the number recruited to the study, and their clinical and demographic characteristics.

B.To determine the proportion of consented patients who develop AKI following cardiac surgery.

C.To measure perioperative changes in MV subgroups and MV associated miRNA, as well as platelet and monocyte activation, and the variance of these measures.

D.To establish protocol adherence, with respect to the adequacy and timing of the blood samples that are taken and the calculation of creatinine clearance perioperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing congenital heart operations with cardio-pulmonary bypass.
2. Patients aged ≤ 17 years of age.
3. Patients with a body weight > 2kg.

Exclusion Criteria:

1. Patients with pre-existing inflammatory state: sepsis undergoing treatment, acute kidney injury within 5 days or chronic inflammatory disease.
2. Emergency (operation before the beginning of the next working day after decision to operate) or salvage procedure (patients requiring cardiopulmonary resuscitation - external cardiac massage - en route to the operating theatre or prior to induction of anaesthesia. This does not include cardiopulmonary resuscitation following induction of anaesthesia)
3. Patients where Extracorporeal Membrane Oxygenation (ECMO) support is required.
4. Patients likely to require ECMO postoperatively.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing cardiac surgery in a tertiary academic cardiac surgery unit
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
change from baseline in annexin V positive microvesicles | Pre-operatively, 6-12 hrs post-op and 24 hrs post-op
  Mean plasma concentration of Annexin V positive MV and the concentration variance in plasma from arterial blood samples collected prior to anaesthetic induction, and at 6-12 and 24 hours postoperatively.
change from baseline in microvesicles derived miRNA | Pre-operatively, 6-12 hrs post-op and 24 hrs post-op
  Mean plasma concentration of MV derived miRNA and the concentration variance in plasma from arterial blood samples collected prior to anaesthetic induction, and at 6-12 and 24 hours postoperatively.

SECONDARY OUTCOMES:
Eligibility | pre-operatively
  Since this is a feasibility study, the investigators will evaluate the rate of patients who are eligible among the whole population of screened patients
Recruitment | preoperatively
  Since this is a feasibility study, the investigators will evaluate the rate of patients who will be recruited among the whole population of approached patients
Protocol non-adherence | Pre-operatively, 6-12 hrs post-op and 24 hrs post-op
  Since this is a feasibility study, the investigators will evaluate protocol non-adherence defined as the failure to obtain the specified blood volume or urine sample required for analysis at the required time.
Acute Kidney Injury | preoperatively, postoperatively every day until day 7
  Acute kidney injury defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Variation in Renal inflammation | Pre-operatively, 6-12 hrs post-op and 24 hrs post-op
  Variation in Renal inflammation will be determined by variation in values of urine Neutrophil Gelatinase-Associated Lipocalin (NGAL) and Liver type- Fatty Acid Binding Protein (L-FABP) and urinary nitric oxide bioavailability .
Incidence of Acute Lung Injury - Low Cardiac Output | preoperatively, postoperatively every day until day 7
  Acute Lung Injury (PaO2/FiO2<300mmHg)
Incidence of Low Cardiac Output | preoperatively, postoperatively every day until day 7
  Low Cardiac Output (the use of two or more inotropes)
Variation in pro-coagulant potential of microvesicles | Pre-operatively, 6-12 hrs post-op and 24 hrs post-op
  This is a measure of MV tissue factor expression and indicates the likely pro-inflammatory effect of the MV.
Variations in sources of microvesicles | Pre-operatively, 6 - 12 hrs post-op and 24 hrs post-op
  Sources of MV: platelet, endothelial and monocyte activation will be determined by flow cytometry.
Variations in systemic inflammatory cytokine response | Pre-operatively, 6 - 12 hrs post-op and 24 hrs post-op
  The systemic inflammatory cytokine response will be quantified by measurement of serum interleukin-8, interleukin-6, tumor necrosis factor -α, monocyte chemotactic protein -1, monocyte chemotactic protein -3, intercellular adhesion molecule, E-selectin.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin J Murphy, Prof, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Sullo N, Mariani S, JnTala M, Kumar T, Wozniak MJ, Smallwood D, Pais P, Westrope C, Lotto A, Murphy GJ. An Observational Cohort Feasibility Study to Identify Microvesicle and Micro-RNA Biomarkers of Acute Kidney Injury Following Pediatric Cardiac Surgery. Pediatr Crit Care Med. 2018 Sep;19(9):816-830. doi: 10.1097/PCC.0000000000001604. PMID 29912813